CLINICAL TRIAL: NCT03385863
Title: A Multicenter Clinical Study on the Comparison of the Efficacy of Surfactant and Perinatal Risk Factors in NRDS With Different Gestational Ages
Brief Title: Efficacy of Surfactant and Perinatal Risk Factors in NRDS With Different Gestational Ages
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Li Wang, Daping Hospital, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: 02333669
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Infant, Newborn, NRDS
MeSH Terms: interventions — Surface-Active Agents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- early preterm infants with RDS: gestational age<34 weeks
  Interventions: Drug: Surfactant, Pulmonary，Curosurf; Other: Perinatal risk factors of NRDS
- near term infants with RDS: 34 weeks≤gestational age< 37 weeks
  Interventions: Drug: Surfactant, Pulmonary，Curosurf; Other: Perinatal risk factors of NRDS
- term infants with RDS: Gestational age ≥ 37 weeks
  Interventions: Drug: Surfactant, Pulmonary，Curosurf; Other: Perinatal risk factors of NRDS

INTERVENTIONS:
Drug: Surfactant, Pulmonary，Curosurf — All NRDS were given an early endotracheal infusion of Curosuf, with an initial dose of 200mg/kg, and if the condition needed to be repeated. Compare the therapeutic effect of pulmonary surfactant of infants at different gestational ages and to investigate whether exogenous surfactant replacement therapy is effective for all newborns with RDS.
Other: Perinatal risk factors of NRDS — Compare the perinatal risk factors that were closely related to NRDS between early preterm infants with RDS and near term/term infants with RDS.

SUMMARY:
Since exogenous surfactant replacement therapy was first used to prevent neonatal respiratory distress syndrome (NRDS)，it has become the main method of treatment of NRDS. However, in some infants, death is inevitable despite intensive care and surfactant replacement therapy, especially in near-term and term infants. The first goal of our study is to compare the therapeutic effect of pulmonary surfactant of infants at different gestational ages and to investigate whether exogenous surfactant replacement therapy is effective for all newborns with RDS. The second goal of our study is to further analyze the risk factors and causes of RDS in early preterm infants and near term/term infants.

ELIGIBILITY:
Inclusion Criteria:

Infants with RDS who received surfactant therapy were recruited between January 2011 and December 2016.

Exclusion Criteria:

Infants were excluded if they had any congeni- tal malformation, inherited metabolic abnormality, intrauterine infection, Rh/Rh incompatibility, pneumonia, pulmonary hypertension, meconium aspiration syndrome, or asphyxia.

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with RDS who received surfactant therapy were recruited from 24 hospitals between January 2011 and December 2016.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
therapeutic effect of pulmonary surfactant of infants at different gestational ages | January 1，2011 to December 30，2016

CONTACTS AND LOCATIONS:
Overall Officials: Li Wang, Doctor, Principal Investigator — Daping Hospital, Third Military Medical University
Locations (1):
- Department of pediatrics, Daping Hospital, The Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided